CLINICAL TRIAL: NCT03635333
Title: Effects of E-Cigarette Flavors on Adults
Brief Title: Effects of E-Cigarette Flavors on Adults TCORS 2.0
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2000023077-2; 2U54DA036151-06 (NIH)
Record Dates: First submitted 2018-08-13; First posted 2018-08-17 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Nicotine Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine; Flavoring Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Low nicotine, tobacco (Experimental): 6 mg nicotine combined with tobacco flavored e-juice
  Interventions: Drug: Nicotine; Drug: Flavor
- Low nicotine, menthol (Experimental): 6 mg nicotine combined with menthol flavored e-juice
  Interventions: Drug: Nicotine; Drug: Flavor
- Low nicotine,cherry (Experimental): 6 mg nicotine combined with cherry flavored e-juice
  Interventions: Drug: Nicotine; Drug: Flavor
- High nicotine, tobacco (Experimental): 18 mg nicotine combined with tobacco flavored e-juice
  Interventions: Drug: Nicotine; Drug: Flavor
- High nicotine, menthol (Experimental): 18 mg nicotine combined with menthol flavored e-juice
  Interventions: Drug: Nicotine; Drug: Flavor
- High Nicotine, cherry (Experimental): 18 mg nicotine combined with cherry flavored e-juice
  Interventions: Drug: Nicotine; Drug: Flavor
- Low Nicotine, Vanilla (Experimental): 6 mg nicotine combined with vanilla flavored e-juice
  Interventions: Drug: Nicotine; Drug: Flavor
- High Nicotine, Vanilla (Experimental): 18 mg nicotine combined with vanilla flavored e-juice
  Interventions: Drug: Nicotine; Drug: Flavor

INTERVENTIONS:
Drug: Nicotine — Nicotine level (6 or 18 mg)
Drug: Flavor — Flavor of e-juice (tobacco, menthol, cherry, vanilla)

SUMMARY:
This study looks at the effects of flavors when administered with nicotine in e-cigarettes in younger and older adult cigarette smokers.

DETAILED DESCRIPTION:
This study looks at the effects of flavors when administered with nicotine in e-cigarettes in younger and older adult cigarette smokers. Regular cigarette smokers who do not want to quit smoking will be asked to complete 3 lab sessions in which they will use an e-cigarette and complete questionnaires. This will be followed by a two-week period where participants are asked to stop using cigarettes and other tobacco products and to only use the e-cigarettes provided. Researchers will examine the influence of flavors (sweet, cool, tobacco) on reward (liking/wanting) from e-cigs containing one of two nicotine concentrations (6 mg/ml, 18 mg/ml) following acute tobacco abstinence.

As of October 2020, this protocol was updated in which an additional lab session was added. Participants are to complete 4 lab sessions in which they will use an e-cigarette and complete questionnaires. In each individual lab session, they will sample one of the following four e-liquids: cherry, vanilla, menthol, tobacco. Additionally, participant age range was shifted to 21-50 with the younger condition being 21-34 and older being 35-50 and cigarette requirement was at least 1 cigarette/day at this time to be more representative of current persons who smoke.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21-34 years or 35 -50 years
* Able to read and write
* Smoking >/= 1 cigarettes or cigars/day
* Willing to abstain from regular smoking for 2 weeks and use only e-cigarettes
* Not seeking treatment to stop smoking

Exclusion Criteria:

* Daily use of other drugs including prescribed psychoactive drugs
* Any significant current medical or psychiatric condition
* Known hypersensitivity to propylene glycol
* Pregnant or lactating females

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CMHC, Substance Abuse Center, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- High Nicotine: 18 mg nicotine
- Low Nicotine: 6mg/ml nicotine
Period: Overall Study
Arm/Group | High Nicotine | Low Nicotine
Started | 63 | 67
Vanilla Flavor | 52 | 55
Cherry Flavor | 51 | 51
Menthol Flavor | 57 | 59
Tobacco Flavor | 56 | 59
Completed | 58 | 56
Not Completed | 5 | 11

BASELINE CHARACTERISTICS:
Population: Participants included in the primary analyses (those who were enrolled in the updated study design October 2020).
Groups:
- Low Nicotine Group (6mg/ml): Participants that were assigned to the low nicotine condition and exposed to tobacco, menthol, cherry, and vanilla.
- High Nicotine Group (18mg/ml): Participants that were assigned to the high nicotine condition and exposed to tobacco, menthol, cherry, and vanilla.
- Total: Total of all reporting groups
Arm/Group | Low Nicotine Group (6mg/ml) | High Nicotine Group (18mg/ml) | Total
Number analyzed (Participants) | 62 | 59 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (8.8) | 35.8 (7.5) | 35.9 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 21 | 46
  Male | 37 | 38 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 4 | 13
  Not Hispanic or Latino | 53 | 55 | 108
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 10 | 20
  White | 42 | 37 | 79
  More than one race | 4 | 4 | 8
  Unknown or Not Reported | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 62 | 59 | 121

OUTCOME MEASURES:

1. Primary Outcome: Change Score in Liking/Wanting of E-cigarette
Description: The Labeled Hedonic Scale (LHS; Lim et al., 2009) will be used to ask about liking and wanting of the e-cigarette (one item VAS scale [range -100 to 100] with ratings from most disliked sensation imaginable to most liked sensation imaginable with higher values indicating greater liking)
Time Frame: Baseline (+10 minutes) to end of lab session (+40 minutes)
Population: The study started in May 2019 and the study was active between May 2019 and October 2020 and 9 participants were enrolled. However, due to study changes communicated previously, analyses only reflect enrolled participants who completed the study following the study protocol change (i.e., addition of a laboratory session in October 2020). Randomized non-starters were excluded from analyses (n=8, 5 low nicotine, 3 high nicotine). Those who completed at least one lab had data included in analyses
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Low Nicotine, Tobacco | Low Nicotine, Menthol | Low Nicotine,Cherry | High Nicotine, Tobacco | High Nicotine, Menthol | High Nicotine, Cherry | Low Nicotine, Vanilla | High Nicotine, Vanilla
Number analyzed (Participants) | 53 | 53 | 53 | 54 | 54 | 55 | 52 | 53
units on scale | -1.06 (4.68) | -5.59 (4.67) | -7.14 (4.8) | -7.63 (4.72) | 8.41 (4.73) | 0.42 (4.78) | 4.77 (4.65) | 5.48 (4.74)

ADVERSE EVENTS:
Time Frame: Adverse events for each participant were recorded from the start of their participant to completion (6 month follow up phone call), on average 6 months.
Groups:
- Vanilla Low Nicotine Group (6mg/ml): Participants who were assigned to the low nicotine condition and were exposed to vanilla flavor.
- Vanilla High Nicotine Group (18mg/ml): Participants who were assigned to the high nicotine condition and were exposed to vanilla flavor.
- Cherry Low Nicotine Group (6mg/ml): Participants who were assigned to the low nicotine condition and were exposed to cherry flavor.
- Cherry High Nicotine Group (18mg/ml): Participants who were assigned to the high nicotine condition and were exposed to cherry flavor.
- Tobacco Low Nicotine Group (6mg/ml): Participants who were assigned to the low nicotine condition and were exposed to tobacco flavor.
- Tobacco High Nicotine Group (18mg/ml): Participants who were assigned to the high nicotine condition and were exposed to tobacco flavor.
- Menthol Low Nicotine Group (6mg/ml): Participants who were assigned to the low nicotine condition and were exposed to menthol flavor.
- Menthol High Nicotine Group (18mg/ml): Participants who were assigned to the high nicotine condition and were exposed to menthol flavor.
- Randomized Non-Starter Low Nicotine Group (6mg/ml): Participants who were randomized to the low nicotine condition and enrolled in the trial but did not start lab and thus had no flavor exposure
- Randomized Non-starter High Nicotine Group (18mg/ml): Participants who were randomized to the high nicotine condition and enrolled in the trial but did not start lab and thus had no flavor exposure
Arm/Group | Vanilla Low Nicotine Group (6mg/ml) | Vanilla High Nicotine Group (18mg/ml) | Cherry Low Nicotine Group (6mg/ml) | Cherry High Nicotine Group (18mg/ml) | Tobacco Low Nicotine Group (6mg/ml) | Tobacco High Nicotine Group (18mg/ml) | Menthol Low Nicotine Group (6mg/ml) | Menthol High Nicotine Group (18mg/ml) | Randomized Non-Starter Low Nicotine Group (6mg/ml) | Randomized Non-starter High Nicotine Group (18mg/ml)
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/52 | 0/51 | 0/51 | 0/59 | 0/57 | 0/59 | 0/56 | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/52 | 0/51 | 0/51 | 0/59 | 0/57 | 0/59 | 0/56 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 0/55 | 0/52 | 1/51 | 0/51 | 1/59 | 0/57 | 0/59 | 0/56 | 0/8 | 0/6
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vanilla Low Nicotine Group (6mg/ml) (N=55) | Vanilla High Nicotine Group (18mg/ml) (N=52) | Cherry Low Nicotine Group (6mg/ml) (N=51) | Cherry High Nicotine Group (18mg/ml) (N=51) | Tobacco Low Nicotine Group (6mg/ml) (N=59) | Tobacco High Nicotine Group (18mg/ml) (N=57) | Menthol Low Nicotine Group (6mg/ml) (N=59) | Menthol High Nicotine Group (18mg/ml) (N=56) | Randomized Non-Starter Low Nicotine Group (6mg/ml) (N=8) | Randomized Non-starter High Nicotine Group (18mg/ml) (N=6)
Other (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Participant stepped on nail between Lab 1 and Lab 2. Participant was treated with antibiotics.
Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Participant reported minor throat irritation from e-cigarette

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/33/NCT03635333/Prot_SAP_001.pdf
  • Informed Consent Form (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/33/NCT03635333/ICF_000.pdf